CLINICAL TRIAL: NCT07034755
Title: Phase II Clinical Study on the Safety and Efficacy of Combined CAR-T Therapy Following Autologous Stem Cell Transplantation in Multiple Myeloma
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Affiliated Hospital of Xuzhou Medical University (Other)
Collaborators: Shuyang People's Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYYY-LL-202502
Record Dates: First submitted 2025-05-17; First posted 2025-06-24 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-05

CONDITIONS: Multiple Myeloma (MM); Allogeneic Hematopoietic Stem Cell Transplantation (HSCT); Chimeric Antigen Receptor T-cell
Keywords: Chimeric Antigen Receptor T-Cell; allogeneic Hematopoietic Stem Cell Transplantation (HSCT); multiple myeloma (MM)
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- The efficacy of autologous hematopoietic stem cell transplantation (ASCT) followed by CAR-T therapy (Experimental): This study evaluates the efficacy and safety of sequential autologous hematopoietic stem cell transplantation (auto-HSCT) followed by CAR-T cell therapy in newly diagnosed multiple myeloma (MM) patients who achieved partial response (PR) or better but failed to attain complete response (CR) after four cycles of first-line chemotherapy, or those who achieved CR but harbored high-risk factors. The clinical data from this research will provide supportive evidence for novel therapeutic strategies in this subset of MM patients.
  Interventions: Other: autologous hematopoietic stem cell transplantation (ASCT) followed by CAR-T therapy

INTERVENTIONS:
Other: autologous hematopoietic stem cell transplantation (ASCT) followed by CAR-T therapy — The efficacy of autologous hematopoietic stem cell transplantation (ASCT) followed by CAR-T therapy was evaluated in patients with multiple myeloma who either achieved partial response (PR) or better (but not complete response [CR]) after four cycles of first-line chemotherapy, or those who achieved CR but had high-risk factors.

SUMMARY:
Chimeric Antigen Receptor T-Cell (CAR-T) immunotherapy is a rapidly developing novel approach in adoptive immunotherapy for tumors in recent years. Its main characteristic lies in genetically engineering T cells to express tumor antigen-specific receptors, thereby endowing them with targeting capability, cytotoxicity, and persistence. This approach has demonstrated remarkable efficacy in relapsed/refractory hematologic malignancies. Research on multiple myeloma (MM)-specific CAR-T cells has also been progressively conducted with promising outcomes, establishing CAR-T cell therapy as an effective new treatment strategy for MM. Notably, targets such as B-cell maturation antigen (BCMA) and GPRC5D have emerged as prominent therapeutic targets for CAR-T cell therapy.

Therefore, we propose to evaluate the efficacy and safety of sequential CAR-T therapy following autologous hematopoietic stem cell transplantation (ASCT) in newly diagnosed MM patients who achieve partial response (PR) or better after four cycles of first-line chemotherapy but fail to attain complete response (CR), or those who achieve CR but present with high-risk factors. The clinical data from this study will provide evidence-based support for novel treatment strategies in this subset of MM patients.

DETAILED DESCRIPTION:
Multiple myeloma (MM) is a malignant plasma cell disorder characterized by abnormal proliferation of bone marrow plasma cells accompanied by excessive production of monoclonal immunoglobulin or light chains (M-protein). It is frequently associated with multiple osteolytic lesions, hypercalcemia, anemia, and renal impairment. The disease has an incidence rate of 2-3 per 100,000, with a male-to-female ratio of 1.6:1, predominantly affecting individuals over 40 years of age.

Traditional treatments for MM include chemotherapy regimens such as MP (melphalan + prednisone), VAD (vincristine + doxorubicin + dexamethasone), and CTD (cyclophosphamide + thalidomide + dexamethasone), as well as radiotherapy and autologous hematopoietic stem cell transplantation (ASCT). However, these approaches are limited by low induction remission rates and short long-term survival.

In recent years, the introduction of novel agents such as proteasome inhibitors (e.g., bortezomib) and immunomodulatory agents (e.g., lenalidomide) has significantly improved remission rates and reduced chemotherapy-related toxicity, extending the median survival of MM patients from 2-3 years to over 5 years. For transplant-eligible patients, intensive induction therapy followed by ASCT remains the current first-line treatment strategy. For relapsed/refractory MM, next-generation oral proteasome inhibitors (e.g., ixazomib), monoclonal antibodies (e.g., daratumumab), and targeted cellular immunotherapies have demonstrated promising efficacy.

Nevertheless, MM remains incurable, and with each relapse, the likelihood of acquiring high-risk cytogenetic abnormalities increases, leading to escalating treatment resistance. Consequently, subsequent relapses are associated with shorter progression-free survival and post-relapse survival durations. Therefore, there is an urgent need to explore more effective therapeutic strategies to improve outcomes and prolong survival in MM patients with high-risk features or suboptimal depth of response.

The treatment of multiple myeloma (MM) with transplantation has evolved through several stages, including autologous stem cell transplantation (auto-HSCT), allogeneic hematopoietic stem cell transplantation (allo-HSCT), and sequential auto-HSCT followed by allo-HSCT. However, due to factors such as the advanced median age at diagnosis of MM patients, allo-HSCT has not become the first-line treatment for most newly diagnosed MM patients.

The sequential approach-first performing auto-HSCT to reduce tumor burden, followed by reduced-intensity allo-HSCT-has shown conflicting clinical efficacy reports, limiting its widespread adoption. Consequently, auto-HSCT remains the primary treatment modality for transplant-eligible MM patients.

Since its introduction in the early 1980s, auto-HSCT has significantly prolonged overall survival (OS) in MM patients and has been regarded as the preferred treatment for newly diagnosed MM patients aged ≤65 years. However, with the emergence of novel drugs (e.g., proteasome inhibitors, immunomodulators, CD38 monoclonal antibodies), the complete response (CR) rate after 4-6 cycles of induction therapy has reached 20%-40%, raising questions about the necessity of auto-HSCT.

Prospective clinical trials comparing auto-HSCT combined with novel agents versus continuous novel drug therapy have demonstrated that auto-HSCT provides greater progression-free survival (PFS)benefits, reaffirming its critical role in newly diagnosed MM. Even with monoclonal antibody-based induction regimens, auto-HSCT remains a cornerstone of treatment for eligible patients.

In summary, despite advancements in pharmacotherapy, auto-HSCT continues to play an indispensable role in achieving deeper remission and prolonging survival** for transplant-eligible MM patients

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-70 years old
* Expected survival: >12 weeks
* Diagnosis: Multiple myeloma confirmed by physical examination, pathological examination, laboratory tests, and imaging studies
* Post-chemotherapy status:
* Patients who achieved partial response (PR) or better but failed to reach complete response (CR) after four cycles of first-line chemotherapy Patients who achieved CR after four cycles of first-line chemotherapy but have high-risk factors
* Liver function:

  * ALT and AST < 3 times the upper limit of normal
  * Bilirubin < 2.0 mg/dl
* Performance status: Karnofsky Performance Status (KPS) >50%
* Organ function: No severe liver, kidney, or heart diseases
* Stem cell transplantation: Eligible for stem cell transplantation
* Venous access: Able to undergo venous blood sampling without contraindications to leukapheresis
* Informed consent: Capable of understanding and voluntarily signing a written informed consent form

Exclusion Criteria:

* Pregnancy or lactation, or women planning pregnancy within the next 6 months
* Infectious diseases(e.g., HIV, active tuberculosis)
* Active hepatitis B or C infection
* Feasibility assessment showing lymphocyte-targeted transfection rate <10% or insufficient expansion (<5-fold) under CD3/CD28 co-stimulation
* Abnormal vital signs or inability to cooperate with examinations
* Psychiatric/psychological disorders precluding treatment compliance or efficacy evaluation
* Severe allergic constitution or history of severe allergies, especially to IL-2
* Systemic or localized severe infection requiring anti-infective therapy
* Severe autoimmune diseases
* Other conditions deemed unsuitable for inclusion by the investigator

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2028-03-01 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival(PFS):Time between treatment and disease progression or death | Pre-hematopoietic stem cell transplant evaluation、assessed at two weeks, 1 month, 2 months, 3 months, 6 months, and 1 year after CAR-T infusion
  The efficacy of autologous hematopoietic stem cell transplantation (ASCT) followed by CAR-T therapy was evaluated in patients with multiple myeloma who either achieved partial response (PR) or better (but not complete response [CR]) after four cycles of first-line chemotherapy, or those who achieved CR but had high-risk factors.
MRD | Efficacy was re-evaluated at 2 weeks, 1 month, 2 months, 3 months, 6 months and 1 year after CAR-T infusion
  Refers to residual tumor cells or small lesions that still exist in the patient's body after treatment but cannot be detected by imaging methods
OS | Efficacy was re-evaluated at 2 weeks, 1 month, 2 months, 3 months, 6 months and 1 year after CAR-T infusion
  The time from the time the patient receives treatment to the patient's death due to any cause

SECONDARY OUTCOMES:
To assess the safety of transplantation in combination with CAR-T | Efficacy was reassessed at two weeks, 1 month, 2 months, 3 months, 6 months, and 1 year after CAR-T infusion
  1. Detection of CRS-related factors: such as IFN, IL-6, TNF, IL-10, IL-4, CRP, etc
  2. Various laboratory tests: blood routine, coagulation function, blood film observation, liver function, kidney function, electrolytes, blood glucose, cardiac enzymes, T cell subsets, immunoglobulins, etc
  3. Observation of adverse events and serious adverse events.

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No